CLINICAL TRIAL: NCT04434053
Title: Adjustable Gravitational vs. Adjustable Differential Pressure Valves in Patients With Idiopathic Normal Pressure Hydrocephalus. Prospective Randomized Study.
Brief Title: Adjustable Gravitational vs. Adjustable Differential Pressure Valves in iNPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Ondřej Bradáč, M.D., M.Sc., Ph.D., Military University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MilitaryUHP
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: iNPH
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIETHKE M.blue® (Experimental)
  Interventions: Device: MIETHKE M.blue®
- MIETHKE proGAV 2.0® (with SA 2.0®) (Active Comparator)
  Interventions: Device: MIETHKE proGAV 2.0® (with SA 2.0®)

INTERVENTIONS:
Device: MIETHKE M.blue® — The programmable shunt will be adjusted through the MIETHKE M.blue® valve.
  Arms: MIETHKE M.blue®
Device: MIETHKE proGAV 2.0® (with SA 2.0®) — The programmable shunt will be adjusted through the MIETHKE proGAV 2.0® valve that will be implanted together with a shunt-assistant SA 2.0®.
  Arms: MIETHKE proGAV 2.0® (with SA 2.0®)

SUMMARY:
The goal of the study is to verify theoretical benefit of ventriculoperitoneal shunting with MIETHKE M.blue® valve in patients with iNPH. The study is designed to assess walking and balance, urinary function, cognitive performance and quality of life before and after shunting and compare the results between the patients with MIETHKE M.blue® and MIETHKE proGAV 2.0® (with SA 2.0®) valves.

DETAILED DESCRIPTION:
Patients who will be referred to Military University Hospital Prague with suspicion of normal pressure hydrocephalus will be tested by conventional methods to consider implantation of a ventriculo-peritoneal shunt. This testing is performed during hospitalization and includes clinical examination of the patient by a neurosurgeon, neurologist and neuropsychologist including neuropsychological questionnaires or tests - MoCA, AVLT, ROCFT, TMT A + B, Phonemic Verbal Fluency Test (N, K, P), Semantic Fluence Test (animals, vegetables), subtest of battery WAIS III and GDS. Clinical examinations are followed by magnetic resonance imaging. Functional testing of cerebrospinal fluid circulation is initiated on the second day unless another cause of the patient's symptoms (AD, Parkinson's disease, vascular dementia, tumor, obstructive type of hydrocephalus - eg aqueductal stenosis, Blake's pouch cyst etc.) is present. The functional testing will involve lumbar infusion test and subsequent external lumbar drainage (ELD) for 120h, including biochemical analysis of CSF during the ELD. After this time, the objective improvement of the patient's gait with the aid of the Dutch Gait Scale will be evaluated with respect to the subjective evaluation by the patient or family (changes in urinary incontinence / urgency, headaches, etc.). If the diagnosis of normotensive hydrocephalus is confirmed, the patient will be indicated for a VP shunt implantation, which is used for permanent derivation of cerebrospinal fluid into the peritoneal cavity. As a result of cerebrospinal fluid derivation, the clinical condition of most of the patients improves. The operation process described by Michael J. Fritsch (Fritsch et al. 2014) will be modified for various valve types in accordance with the manufacturer's recommendations and assumed conditions for proper valve adjustment. Patients will be randomly implanted with a M.blue® or proGAV 2.0® (with SA 2.0®) valve (Christoph Miethke GmbH & Co. KG) in a randomized manner to form two study groups. The efficacy and safety of the proGAV 2.0® (with SA 2.0®) valve has already been confirmed in a randomized prospective study in patients with idiopathic normotensive hydrocephalus (Lemcke et al. 2013). The theoretical benefit of the M.blue® valve lies in the targeted modification of the cerebrospinal fluid diversion during the active time of a day, when the opening pressure of the valve's gravitational unit is controlled according to the angle between the valve and the horizontal line. The basal opening pressure of the valve that has to be overcome in the supine position is controlled with a fixed differential pressure unit. ProGAV 2.0® is an adjustable differential pressure valve implanted with a shunt-assistant SA 2.0®. The shunt-assistant represents a fixed gravity unit that increases the pressure in the standing position, which must be overcome for the cerebrospinal fluid flow through th shunt. The opening pressure of the valve could be selected according to the patient's height and sex. The basal opening pressure of the valve that must be overcome in the supine position is controlled with an adjustable differential pressure unit that can be adjusted before and after the shunt implantation. In both valves, the opening pressure is the sum of the opening pressures of the gravitational and differential pressure units. The theoretical benefit of the M.blue® valve is the possibility of changing the opening pressure of the gravitational unit regulated according to the position of the head in the space and thus aiming more at the pressure conditions when the valve is not parallel to the horizontal line.

Patients will not be familiar with the type of valve implanted with respect to subjective evaluation of patients during the follow-up. Initial valve settings will be in accordance with the manufacturer's recommendations. Follow-up of the patients will be guided in the usual regime according to the natural history of the disease: at one month of follow-up an outpatient clinical examination by a neurosurgeon, including brain CT scan; at three-months of follow-up an evaluation during a two-day hospitalization including collection of the following questionnaires, brain MRI, clinical examination by a neurosurgeon, neurologist and neuropsychologist and collection of cerebrospinal fluid from the pre-chamber for the biochemical analysis; at six-months an outpatient examination by a neurosurgeon; at one year of follow-up an evaluation during a two-day hospitalization including collection of the following questionnaires, brain MRI, clinical examination by a neurosurgeon, neurologist and neuropsychologist and collection of cerebrospinal fluid from the pre-chamber valve for biochemical analysis; at two-years of follow-up an outpatient clinical examination by neurosurgeon and neuropsychologist including brain CT scan including collection of the following questionnaires and collection of the cerebrospinal fluid from the pre-chamber of the valve for biochemical analysis.

For the purpose of the study, the Dutch Gait scale (gait), UI-SF (incontinence) and MoCA (dementia) will be used to assess the outcome of the shunt operation to monitor the severity and nature of the main symptoms during the follow-up in pre-implant, three months, one year and after two years. The SF-12V2 will be used in a similar mode to monitor the quality of life of the patients. Severity of the symptoms will also be assessed by the Kiefer Scale, which was developed directly to monitor patients with idiopathic normotensive hydrocephalus. Charlson comorbidity index will be used to monitor covariates. All clinical examinations by a neurosurgeon will monitor early and late complications of the short-circuit operation (infection, hemorrhage, overdrainage, underdrainage, shunt malfunction), the number of valve setting changes and their range, unscheduled checks and shunt revisions and other unexpected events.

The expected number of patients who will undergo all examinations after an annual check is 40 (20 and 20).

The expected benefit of the study is in particular to confirm the theoretical assumptions of an adjustable gravitational valve in patients with idiopathic normal pressure hydrocephalus and thus in improvement of the quality and life expectancy of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients (between 60 and 85 years old)
* Clinically suspected Normal Pressure Hydrocephalus (NPH) with at least gait and one other symptom from Hakim-Adams triad (incontinence or dementia)
* maximal initial pressure of 20 cmH2O during lumbar infusion test
* Rout during LIT >9mmHg/ml*min
* at least 15% improvement in Gait scale score after ELD
* Conclusion of neuropsychological examination suggestive of iNPH (based on MoCA, Test of phonemic and verbal fluency, RAVLT, ROCFT, TMT A and B, Subtest of WAIS III, GDS)

Exclusion Criteria:

* Aetiology of hydrocephalus other than idiopathic normal pressure hydrocephalus (secondary normal pressure hydrocephalus - history of meningitis or subarachnoid haemorrhage, obstructive type of hydrocephalus - eg aqueductal stenosis, Blake's pouch cyst)
* Intracranial tumor
* Other neurodegenerative diseases may be present (AD, Parkinson's disease, Lewy body dementia, Progressive supranuclear palsy and cerebrovascular diseases), however have to be mild and evaluated in neurological, neuropsychological examinations and on MRI

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Dutch Gait scale in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | Month 3/Year 1
  The Gait Scale, a useful quantitative measure of gait impairment in NPH patients, is a component of a larger measure developed as part of the Dutch normal pressure hydrocephalus study (Boon et al., 1997). The Gait Scale evaluates various aspects of gait, including walking speed, number of steps, stride length, stance, foot-floor clearance, balance, tandem walking ability, turning ability, and start hesitation in 10m of walking. (Ravdin et al., 2008) The score consists of 3 subcategories and ranges 2-40 points with higher score indicating more severe impairment.
Change in MoCA in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | Month 3/Year 1
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. It was created in 1996 by Ziad Nasreddine in Montreal, Quebec. The MoCA assesses several cognitive domains. Score ranges 0-30 points with lower scores indicating more severely impaired cognitive skills.
Change in ICIQ UI-SF in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | Month 3/Year 1
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity, impact on quality of life (QoL) and simple estimation of a cause of urinary incontinence in men and women. The score ranges 0-21 points with higher score indicating more severe impairment.
Change in Kiefer Score in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | Month 3/Year 1
  The Kiefer is a modified clinical grading tool that measures the severity of the three key symptoms (mental deficits, gait disturbance, incontinence) and two additional minor symptoms (headache and dizziness). The overall score may reach values between 0 and 24, with higher scores indicating more severe impairment
Change in SF12 v 2.0 Health Survey in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | Month 3/Year 1
  The SF-12® V2 Health Survey (SF-12 v2.0) (Ware, Kosinski, Turner-Bowker, & Gandek, 2002) is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. Generic patient-reported outcome (PRO) measures like the SF-12 assess general health and well-being [or health-related quality of life (HRQOL)], including the impact of any and all illnesses on a broad range of functional domains. The SF-12 v2 consists of a subset of 12 items from the SF-36® Health Survey (SF-36) (Ware & Sherbourne, 1992; Ware, Snow, Kosinski, & Gandek, 1993) covering the same eight domains of health outcomes, including physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH).

SECONDARY OUTCOMES:
Postoperative changes in valve settings in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | 1 Year
  Any change in the valve settings postoperatively will be recorded together with a degree of individual changes.
Overdrainage in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | 1 Year
  Headaches, dizziness, subdural effusions on imaging methods (MRI, CT) and any unplanned visits will be recorded. Chronic subdural haematomas will be divided to symptomatic/asymptomatic and number of drainages will be recorded.
Shunt revisions in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | 1 Year
  Any shunt revisions will be recorded together with a cause (malfunction etc.)
Shunt related infections in MIETHKE M.blue® vs. MIETHKE proGAV 2.0® (with SA 2.0®) | 1 Year
  Any shunt related infection will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgical department of the Central Military Hospital, 1st Faculty of Medicine of Charles University, Prague, Czechia